CLINICAL TRIAL: NCT06572384
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of Belimumab Administered Subcutaneously in Adults With Interstitial Lung Disease (ILD) Associated With Connective Tissue Disease (CTD)
Brief Title: A Study of the Efficacy and Safety of Belimumab in Adults With Interstitial Lung Disease Associated With Connective Tissue Disease
Acronym: BEconneCTD-ILD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221672; 2024-513018-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-16; First posted 2024-08-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Lung Diseases, Interstitial
Keywords: Interstitial lung disease; Belimumab; Connective Tissue Disease; Autoimmune disease; Lung Diseases; Lung Diseases, Interstitial; Safety; Efficacy; Monoclonal antibody
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases; Autoimmune Diseases; Lung Diseases | interventions — belimumab

STUDY DESIGN:
Intervention Model Description: This is a two-group parallel study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belimumab (Experimental): Participants will receive belimumab in addition to standard therapy.
  Interventions: Biological: Belimumab
- Placebo (Placebo Comparator): Participants will receive placebo in addition to standard therapy.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Belimumab — Belimumab will be administered.
  Other Names: BENLYSTA, GSK1550188
  Arms: Belimumab
Other: Placebo — Placebo will be administered.
  Arms: Placebo

SUMMARY:
Interstitial lung disease (ILD) is a lung condition resulting in inflammation and stiffening of the lung, often associated with connective tissue diseases (CTDs). ILD causes reduction in lung volume, shortness of breath, cough and fatigue therefore has high impact on quality of life and is also the leading cause of death in participants with these conditions. The study will assess whether treatment of CTD-ILD participants with belimumab in addition to standard therapy will result in the stabilization and/or improvement of lung function and improve symptoms associated with ILD with an acceptable safety profile.

ELIGIBILITY:
Inclusion criteria:

* Participants with persistent/worsening active inflammatory disease who have failed to achieve their treatment goal, i. e., those who have experience lack of expected treatment benefit (clinically meaningful improvement in FVC), fail to demonstrate sustained lung function stability or continue to experience worsening of ILD despite initiation of standard therapy or failed to tolerate standard therapy.
* Documented diagnosis of rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), idiopathic inflammatory myopathy (IIM; including polymyositis, dermatomyositis, anti-synthetase syndrome), Sjogren's syndrome (pSS), or mixed connective tissue disease (MCTD) in accordance with internationally recognized classification criteria
* Diagnosis of inflammatory and/or fibrotic ILD on High Resolution Computed Tomography (HRCT) with a total disease extent of greater than or equal to (≥) 10% of the whole lung
* Evidence of persistent active/worsening ILD
* Must be currently receiving stable standard therapy to manage ILD and/or underlying CTD, or to have failed or failed to tolerate standard therapy.
* Participant is capable and willing to self-administer the study medication or has a caregiver who is capable and willing to administer the study medication throughout the study
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

  * Is a woman of nonchildbearing potential (WONCBP) OR
  * Is a Woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of less than (<)1%
* Capable of giving signed informed consent

Exclusion Criteria:

* Diagnosis of ILD other than CTD-ILD.
* Primary diagnosis of Systemic Sclerosis (SSc).
* Participants with rapidly progressive disease (absolute drop of 10% or more of FVC between screening and baseline visit and/or recent pulmonary hospitalization).
* FVC ≤ 45% of predicted, or a Diffusing Capacity of the lung for Carbon Monoxide (DLco) (corrected for hemoglobin) ≤ 40% of predicted at screening as confirmed by central reader
* History or presence of diffuse alveolar hemorrhage (DAH) or other confounding pulmonary disease, signs, or symptoms
* Pulmonary arterial hypertension requiring therapy, as determined by the investigator at, or prior to first day of dosing (Day 1)
* Dependence on continuous oxygen supplementation
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data
* Obstructive pulmonary disease (pre-bronchodilator Forced Expiratory Volume (FEV1) /FVC <0.7) as confirmed by central reader
* Significant emphysema on screening or historical HRCT (extent of emphysema exceeds extent of ILD) as confirmed by central reader
* Confirmed Progressive multifocal leukoencephalopathy (PML) or unexplained new-onset or deteriorating neurologic signs and symptoms
* Participants with patient health questionnaire (PHQ-9) score ≥10, that in the opinion of a mental healthcare professional pose a serious suicide risk, have or any history of suicidal behavior in the last 6 months and/or any suicidal ideation in the last 2 months, or who in the investigator's judgment, poses a significant suicide risk.
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Breast cancer within the past 10 years
* Major surgery (including joint surgery) within 3 months prior to screening or planned during the duration of the study
* An active infection, or a history of infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2028-10-18 (Estimated); Study Completion 2028-12-13 (Estimated)

PRIMARY OUTCOMES:
Absolute Change from Baseline in Forced Vital Capacity (FVC) milliliter (mL) at Week 52 | Baseline and Week 52
  Forced vital capacity is the total amount of air exhaled during the lung function test. Low FVC (mL) reflects more impaired lung function. Absolute Change from Baseline in FVC will be reported.

SECONDARY OUTCOMES:
Absolute Change from Baseline in FVC Percentage (%) Predicted at Week 52 | Baseline and Week 52
  FVC are expressed as a percentage of the predicted normal for a person of the same sex, age, and height. Lower % predicted FVC (mL) reflects more impaired lung function.
Time to ILD Progression or Death | From the date of assignment (Day 1) until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 52 Weeks
  Time taken for a participant to experience ILD progression or death.
Absolute Change from Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue Score at Week 52 | Baseline and Week 52
  The FACIT-Fatigue is a short, 13-item questionnaire that assesses self-reported fatigue and its associated impact for daily activities over the past 7 days. The scale range is from 0 to 52, with 0 being the worst possible score and 52 being the best possible score (indicating less/no fatigue).
Absolute Change from Baseline in Living with Pulmonary Fibrosis (L-PF) Total Symptom Score at Week 52 | Baseline and Week 52
  The L-PF questionnaire is a 49-item questionnaire with two modules: 1) symptoms (28 items) and 2) impacts (21 items). The Symptoms module yields three domain scores: 1) dyspnea, 2) cough and 3) fatigue as well as a total Symptoms score. Participants rate the severity of their symptoms in the last 24 hour on a 5-point rating scale. Scoring is performed as a summary score, the mean of the dimension ratings multiplied by 100. Summary scores range from 0-100, with the higher the score the greater the impairment.
Absolute Change from Baseline in Quantitative Interstitial Lung Disease in the Whole Lung (QILD-WL) At Week 52 | Baseline and Week 52
  Change from baseline in extent of architectural distortion (fibrosis), ground glass opacification, and honeycombing features on High-resolution computed tomography (HRCT) as measured by computer-aided analysis tools. Extent of ILD is calculated by summing pixel counts and expressing this as a percentage of the whole lung. ILD extent can range from 0-100% with higher percentage representing more extensive ILD.
Absolute Change from Baseline in Quantitative Measures of Lung Fibrosis (QLF) in the Whole Lung At Week 52 | Baseline and Week 52
  Change from baseline in extent of reticular patterns with architectural distortion (fibrosis) on HRCT as measured by computer-aided analysis tools. Extent of fibrosis is calculated by summing pixel counts and expressing this as a percentage of the whole lung. Fibrosis extent can range from 0-100% with higher percentage representing more extensive fibrosis.
Absolute Change from Baseline in Quantitative Ground Glass Opacity in the Whole Lung (QGGO-WL) at Week 52 | Baseline and Week 52
  Change from baseline in extent of ground glass opacification (GGO) on HRCT as measured by computer-aided analysis tools. Extent of GGO is calculated by summing pixel counts and expressing this as a percentage of the whole lung. GGO extent can range from 0-100% with higher percentage representing more extensive GGO.
Achieving Relative Decline from Baseline in FVC (mL) ≥ 5% at Week 52 | Baseline and Week 52
Achieving Relative Decline from Baseline in FVC (mL) ≥ 10% at Week 52 | Baseline and Week 52
Absolute Change from Baseline in Steroid Dose (Prednisone Equivalent Dose) at Week 52 | Baseline and Week 52
Time to Connective Tissue Disease Progression | Up to 52 Weeks
  Time taken for a participant to experience CTD progression.
Absolute Change from Baseline in Transition Dyspnea Index (TDI) at Week 52 | Baseline and Week 52
  TDI assess dyspnea severity at baseline and its change over time. TDI includes 3 components: functional impairment, magnitude of task and magnitude of effort. Each component has 7 grades, ranging from -3 (major deterioration) to +3 (major improvement), which are summed to calculate a score, ranging between - 9 and +9. Lower score indicates more severely the participant is affected by dyspnea.
Absolute Change from Baseline in Short Form Health Survey 36-Item Version 2 (SF36-v2) at Week 52 | Baseline and Week 52
  The SF-36 yields an 8-scale profile of functional health and well-being scores as well as physical and mental component health summary scores. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score (0) the more disability.
Absolute Change from Baseline in Living with Pulmonary Fibrosis (L-PF) Impacts Total Score at Week 52 | Baseline and Week 52
  The L-PF questionnaire is a 49-item questionnaire with two modules: 1) symptoms (28 items) and 2) impacts (21 items). The Symptoms module yields three domain scores: 1) dyspnea, 2) cough and 3) fatigue as well as a total Symptoms score. Participants rate the severity of their symptoms in the last 24 hour on a 5-point rating scale. Scoring is performed as a summary score, the mean of the dimension ratings multiplied by 100. Summary scores range from 0-100, with the higher the score (100) the greater the impairment.
Absolute Change from Baseline in King's Brief Interstitial Lung Disease Questionnaire (K-BILD) at Week 52 | Baseline and Week 52
  The K-BILD questionnaire consists of 15 items (assessed by the participants on a scale ranging from 1 to 7, where 1 and 7 represent worst and best health status). Items are compiled into 3 domains: breathlessness and activities (range: 0-21), psychological (range: 0-34), and chest symptoms (range: 0-8). Scores are transformed to a range of 0-100 by using logit values (higher scores indicate better health status). A total score and 3 domain scores are calculated ranging from 0-100 with greater scores (100) denoting better quality of life.
Absolute Change from Baseline in Physician Global Assessment (PhGA) at Week 52 | Baseline and Week 52
  The PhGA is a score which enables the treating physician to rate the participants disease on a scale from 0 to 10, where higher score (10) indicates greater severity.
Absolute Change in Patient Global Impression of Change (PGIC)-ILD at Week 52 | Baseline and Week 52
  The PGIC contains two items, a global question asking participants to rate their overall change in ILD severity since first starting this study using a 7-point verbal rating scale, and a yes/no question asking participants to indicate whether the change is meaningful from their perspective.
Absolute Change from Baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLco) % Predicted at Week 52 | Baseline and Week 52
Number of Participants with Adverse Events (AEs), Adverse Events of Special Interest (AESIs) Serious Adverse Events (SAEs) | Up to Week 60
Number of Participants with Respiratory Related Hospitalizations up to Week 52 | Up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (102):
- United States (13):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Potsdam, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Salt Lake City, Utah
- Argentina (7):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Santa Fe
- Australia (3):
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Spearwood, Western Australia
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Namur
- Brazil (5):
  - GSK Investigational Site, Barra Mansa
  - GSK Investigational Site, Juiz de Fora
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São José do Rio Preto
  - GSK Investigational Site, São Paulo
- Canada (2):
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- China (12):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Mianyang
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Nanning
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Suzhou
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Zhuzhou
- France (6):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Pessac
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Toulouse
- Germany (4):
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Minden
  - GSK Investigational Site, Würzburg
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Larissa
- Italy (10):
  - GSK Investigational Site, Ancona
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Modena
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Pisa
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Udine
  - GSK Investigational Site, Verona
- Japan (11):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Miyazaki
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Yamanashi
- Mexico (5):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexicali
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Mérida
- Netherlands (3):
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- GSK Investigational Site, Panama City, Panama
- South Korea (4):
  - GSK Investigational Site, Bucheon Kyunggi-Do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Kyunggi-do
  - GSK Investigational Site, Yongsan-Ku Seoul
- Spain (8):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- United Kingdom (3):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/